CLINICAL TRIAL: NCT00272740
Title: An Open, Multicenter Phase II Trial Evaluating the Antitumour Efficacy of Faslodex® (Fulvestrant) in Postmenopausal Women With Advanced Breast Cancer Failing Non-Steroidal or Steroidal Aromatase Inhibitors
Brief Title: SAKK - a Trial to Evaluate Antitumor Efficacy of Faslodex® After Aromatase Inhibitor Failure in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9238SZ/0001; SAKK; 21/00
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2007-02-09 (Estimated); Status verified 2007-02

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; fulvestrant; Faslodex; hormonotherapy; aromatase inhibitor failure; Advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant

SUMMARY:
The primary objective of the study is to assess the activity of fulvestrant in postmenopausal women with advanced breast cancer failing treatment with non-steroidal or steroidal aromatase inhibitors by estimating the Clinical Benefit Rate

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmation of breast cancer
* progression under treatment with an aromatase inhibitor
* At least one measurable or non-measurable lesion

Exclusion Criteria:

* Prior treatment for breast cancer with more than 2 different hormonal agents
* More than 1 chemotherapy for advanced disease
* Presence of life-threatening metastatic visceral disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93
Dates: Start 2000-03

PRIMARY OUTCOMES:
Clinical Benefit Rate

SECONDARY OUTCOMES:
Duration of clinical benefit
Time to progression
Duration of response
Time to treatment failure
Safety and tolerability
6. clinical benefit rate according to HER2/neu status

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Switzerland Medical Director, MD, Study Director — AstraZeneca
Locations (8):
- Research Site, Leuven, Belgium
- Switzerland (7):
  - Research Site, Aarau
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Mendrisio
  - Research Site, Milano
  - Research Site, Sankt Gallen